CLINICAL TRIAL: NCT03333824
Title: A Phase I Open-label Study to Evaluate the Effect of Multiple Doses of AZD1775 on the Pharmacokinetics of Substrates for CYP3A, CYP2C19, CYP1A2 and to Provide Data on the Effect of AZD1775 on QT Interval in Patients With Advanced Solid Tumours
Brief Title: Effects of AZD1775 on the PK Substrates for CYP3A, CYP2C19, CYP1A2 and on QT Interval in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6014C00006
Record Dates: First submitted 2017-10-23; First posted 2017-11-07 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Solid Tumours
Keywords: Pharmacokinetics, Cardiac Conduction, Mitotic Checkpoint inhibitor, QTc interval
MeSH Terms: interventions — Cytochrome P-450 CYP1A2; Caffeine; Cytochrome P-450 CYP2C19; Omeprazole; Cytochrome P-450 CYP3A; Midazolam; Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Wee-1 kinase inhibitor AZD1775 (Experimental): To evaluate the effect of multiple doses of AZD1775 on the PK of substrates for CYP3A (midazolam), CYP2C19 (omeprazole), CYP1A2 (caffeine) and to evaluate the effect of multiple doses of AZD1775 on QT interval
  Interventions: Drug: CYP1A2 (caffeine); Drug: CYP2C19 (omeprazole); Drug: CYP3A (midazolam); Drug: Kytril (granisetron); Drug: Wee-1 kinase inhibitor AZD1775

INTERVENTIONS:
Drug: CYP1A2 (caffeine) — In Part A, Period 1, patients will be administered a 3 drug cocktail of caffeine, omeprazole and midazolam on Day -8 followed by a washout period of at least 7 but no more than 14 days. In Part A, Period 2, AZD1775 capsules will be administered orally, 225 mg bid, until steady state for 2.5 days (total of 5 doses) and administered together with the cocktail on the morning of Day 3.
Drug: CYP2C19 (omeprazole) — In Part A, Period 1, patients will be administered a 3 drug cocktail of caffeine, omeprazole and midazolam on Day -8 followed by a washout period of at least 7 but no more than 14 days. In Part A, Period 2, AZD1775 capsules will be administered orally, 225 mg bid, until steady state for 2.5 days (total of 5 doses) and administered together with the cocktail on the morning of Day 3.
Drug: CYP3A (midazolam) — In Part A, Period 1, patients will be administered a 3 drug cocktail of caffeine, omeprazole and midazolam on Day -8 followed by a washout period of at least 7 but no more than 14 days. In Part A, Period 2, AZD1775 capsules will be administered orally, 225 mg bid, until steady state for 2.5 days (total of 5 doses) and administered together with the cocktail on the morning of Day 3.
Drug: Kytril (granisetron) — Patients should be administered Kytril (granisetron) 1 mg orally, under fasted conditions (-2 to 2 hours away from meals), 30 minutes prior to administration of the AZD1775 capsules with a small amount of water.
Drug: Wee-1 kinase inhibitor AZD1775 — Multiple doses of 225 mg AZD1775, (3 x 75 mg, printed capsules) administered orally. The drug class of AZD1775 is Wee-1 kinase inhibitor.

SUMMARY:
The purpose of this study is to determine whether AZD1775 has any effect on the pharmacokinetics (PK) of three compounds (caffeine, omeprazole, and midazolam) that are probes for common drug-metabolizing enzymes (caffeine-CYP1A2, omeprazole-CYP2C19, midazolam-CYP3A). The study also seeks to determine the effect of AZD1775 on the QTc interval, which is a common measure of cardiac (heart) function.

DETAILED DESCRIPTION:
This is a Phase I, 2-part study (Part A and Part B) in patients with advanced solid tumours.

Part A: Part A of this study is an open-label, non-randomised, 2-period design. The treatment starts with the administration of a cocktail of 3 medications:

caffeine, omeprazole and midazolam (Day -8), followed by pharmacokinetic (PK) sampling for 24 hours (Period 1) and a washout period of at least 7, but no more than 14 days. In Period 2, AZD1775 will be administered twice daily (bid) until steady state for 2.5 days (total of 5 doses) and the final dose will be administered in combination with the cocktail in the morning of Day 3.

Part B: Part B is an open-label, non-randomised study in the same patients who participated in Part A. On Day -1, baseline dECG assessments will be performed at clock times matched to planned/scheduled dECG assessment times on Days 1 and 3.

Starting on Day 1, each patient will receive AZD1775 (225 mg) bid for 2.5 days and will undergo dECG and PK assessments pre-dose and for 12 hours post AZD1775 dose.

On Day 3, patients will receive their final AZD1775 dose and undergo dECG and PK assessments pre-dose and for 12 hours post-dose. On completion of Part B (ie, collection of the 24-hour PK sample/dECG and safety assessments on Day 4) patients will enter a 4-day washout period relative to the last dose of AZD1775. Within 3 days after the washout period, patients will be required to attend an end of treatment (EoT) visit. Patients will be evaluated for their eligibility and interest to enrol into the open-label continued access (CA) study (D6014C00007).

ELIGIBILITY:
Inclusion Criteria:

* Has read and understands the informed consent form (ICF) and has given written informed consent prior to any study procedures.
* Histologically or cytologically documented, locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
* Any prior palliative radiation must have been completed at least 7 days prior to the start of study treatment (first administration of cocktail [Part A Day -8]), and patients must have recovered from any acute adverse effects prior to the start of study treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 1.
* Baseline laboratory values within 7 days of study treatment initiation (first administration of cocktail [Part A Day -8]):

  * Absolute neutrophil count (ANC) ≥1500/μL.
  * Haemoglobin ≥9 g/dL.
  * Platelets ≥100,000/μL.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if known hepatic metastases.
  * Serum bilirubin within normal limits (WNL) or ≤1.5 x ULN in patients with liver metastases; or total bilirubin ≤3.0 x ULN with direct bilirubin WNL in patients with well documented Gilbert's Syndrome.
  * Serum creatinine ≤1.5 x ULN, or measured creatinine clearance (CrCl) calculated by Cockcroft-Gault method ≥45 mL/min (confirmation of creatinine clearance is only required when creatinine is >1.5 x ULN).

CrCl (glomerular filtration rate) = (140-age) x (weight/kg) x F (72 x serum creatinine mg/dL)

awhere F = 0.85 for females and F = 1 for males

* Female patients who are not of childbearing potential and fertile females of childbearing potential who agree to use adequate contraceptive measures that are in place during screening (or consent), for the duration of the study, and for 1 month after treatment stops, and who are not breastfeeding, and who have a negative serum or urine pregnancy test prior to the start of study treatment (first administration of cocktail [Part A Day -8]). Any patient taking an oral contraceptive must be discussed with the Medical Monitor to ensure that there will be no interaction with the brand of oral contraceptive and cocktail of drugs prior to trial entry to confirm eligibility.
* Male patients should be willing to use barrier contraception (ie, condoms) for the duration of the study and for 3 months after study treatment discontinuation.
* Female and/or male patients ≥18 years of age.
* Willingness and ability to comply with the study and follow-up procedures.

For inclusion in the optional genetic component of the study for all the patients:

o Provision of informed consent for genetic research. If a patient declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study, as long as all the eligibility criteria are met.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca personnel and/or personnel at the study centre).
* Previous enrolment or randomisation and received study treatment in the present study. Patients can, however, be re-screened if the reason for the screen failure no longer exists.
* Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or haemorrhage for at least 2 weeks after treatment (including brain radiotherapy). Must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrolment.
* Use of any anti-cancer treatment drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of AZD1775. For drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the prior treatment and administration of AZD1775 treatment is required.
* No other anticancer-therapy (chemotherapy, immunotherapy, hormonal anti-cancer therapy, radiotherapy [except for palliative local radiotherapy]), biological therapy or other novel agent is to be permitted while patient is receiving study treatment. Patients on LHRH analogue treatment for more than 6 months are allowed entry into the study and may continue at the discretion of the Investigator.
* Previous radiation therapy completed ≤7 days prior to the start of study treatment (i.e., first administration of cocktail [Part A Day -8]).
* Major surgical procedures ≤28 days of beginning study treatment (i.e., first administration of cocktail [Part A Day -8]), or minor surgical procedures ≤7 days. No waiting period required following port-a-cath placement or other central venous access placement.
* Grade >1 toxicities from previous cancer therapy, according to the Common Terminology Criteria for Adverse Events [CTCAE]), excluding alopecia or anorexia.
* Patient has an inability to swallow oral medications. Note: Patient may not have a percutaneous endoscopic gastrostomy tube or be receiving total parenteral nutrition.
* Patients suffering from conditions which are likely to adversely affect gastrointestinal motility and/or transit (for example, diarrhoea, vomiting or nausea, gastroparesis, irritable bowel syndrome and malabsorption), or patients with gastrointestinal resection (e.g., partial or total gastrectomy) likely to interfere with absorption of study treatment).
* Patients who are not non-smokers or light smokers (no more than 5 cigarettes per day) and who cannot abstain from smoking from 2 weeks prior to first dose of cocktail until after the last PK sample collection in Part B.
* Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the start of treatment (i.e., first administration of cocktail [Part A Day -8]).
* Excessive intake of caffeine (more than 6 cups of coffee or equivalent per day) and/or consumption of any caffeine containing drinks or food, e.g., coffee, tea, chocolate, caffeine-containing energy drinks (e.g., Red Bull), or cola within 36 hours of administration of the cocktail on Day -8.
* Patient has had prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, which cannot be discontinued 2 weeks prior to the first administration of AZD1775 (Part A Day 1), or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to beginning study treatment (i.e., first administration of cocktail [Part A Day -8]) and withheld throughout the study until 2 weeks after the last administration of AZD1775. Co-administration of aprepitant or fosaprepitant during this study is prohibited. Any patient taking an oral contraceptive must be discussed with the Medical Monitor to ensure that there will be no interaction with the brand of oral contraceptive and cocktail of drugs prior to trial entry to confirm eligibility.
* Patient has had prescription or non-prescription drugs or other products known to be moderate to strong inhibitors/inducers of CYP1A2 or CYP2C19 which cannot be discontinued 2 weeks prior to beginning study treatment (ie, first administration of cocktail [Part A Day -8]) and withheld through Day 4 of Part A
* Patient has had adjustments to prescription or non-prescription drugs or other products known to be mild inhibitors and/or inducers of CYP3A4 within 1 week prior to the first dose of the cocktail (Part A Day -8).
* Herbal preparations taken within 7 days beginning study treatment (i.e., first administration of cocktail [Part A Day -8]). However, in the case of St John's wort, patients cannot have taken this herbal preparation 21 days prior to first dose of cocktail (Part A Day -8). In the case of Angelica root (Bhai Zhi), patients cannot have taken this herbal preparation 2 weeks prior to beginning study treatment (ie, first administration of cocktail [Part A Day -8]).
* Patients taking any concomitant medications that might affect QT/QTc intervals.
* Patients who have taken any proton pump inhibitors (omeprazole, lansoprazole, esomeprazole, pantoprazole, etc.) within 7 days of beginning study treatment (i.e., first administration of cocktail [Part A Day -8]).
* Patients who cannot withhold antacids for 6 hours or H2-antagonists (cimetidine, ranitidine, famotidine, nizatidine) for up to 96 hours at a time (24 hours prior to and following cocktail administration and 24 hours prior to and following AZD1775 administration) .
* Patients who have received midazolam and/or omeprazole (or esomeprazole) within 14 days of beginning study treatment (i.e., first administration of cocktail [Part A Day -8]).
* Any known hypersensitivity or contraindication to the cocktail drugs (caffeine, omeprazole and midazolam) or AZD1775, or to the components thereof.
* Any of the following cardio-vascular conditions currently or within the last 6 months:

  * Unstable angina pectoris.
  * Congestive heart failure ≥ Class 2 as defined by the New York Heart Association
  * Acute myocardial infarction.
  * Significant conduction abnormalities, e.g., atrioventricular block II and III, sick sinus syndrome even if controlled with medication, as well as complete left bundle branch block (complete LBBB).
  * Ventricular or supraventricular arrhythmias.
  * Insufficiently controlled hypertension, i.e., >160/100 mm Hg.
  * Cardiac devices (pacemaker, implantable cardioverter defibrillator, cardiac resynchronisation therapy device, etc.) that can affect the ST-T wave morphology and has a subsequent negative impact on the accuracy of the QTc measurement
* Patients with centrally reviewed QT interval (specifically QTc calculated using the Fridericia formula) >450 ms [QTcF]) obtained from 3 dECGs 2 to 5 minutes apart at study entry, or congenital long QT syndrome.
* AZD1775 should not be given to patients who have a history of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected. AZD1775 has not been studied in patients with ventricular arrhythmias or recent myocardial infarction.
* Pregnant or lactating female patients.
* Serious, symptomatic active infection at the time of study entry, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment.
* Presence of other active invasive cancers.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Active infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).

Any of the following is regarded as a criterion for exclusion from the optional pharmacogenetic part of the study:

* Previous bone marrow transplant.
* Non-leukocyte depleted whole blood product within 120 days of the genetic sample collection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Part A: Area under the plasma concentration-time curve from zero to infinity for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8 and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post cocktail dose
  To assess the effect of AZD1775 on the PK of probe substrates for CYP1A2 (caffeine), CYP2C19 (omeprazole), and CYP3A (midazolam)
Part A: Area under the plasma concentration-time curve from time zero to the time "t" of the last quantifiable concentration for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8 and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post cocktail dose
  To assess the effect of AZD1775 on the PK of probe substrates for CYP1A2 (caffeine), CYP2C19 (omeprazole), and CYP3A (midazolam)
Part A: maximum plasma drug concentration for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8 and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post cocktail dose
  To assess the effect of AZD1775 on the PK of probe substrates for CYP1A2 (caffeine), CYP2C19 (omeprazole), and CYP3A (midazolam)
Part B: dECG intervals (QTcF) for absolute values and time-matched change from baseline | dECGs are measured on Day -1, Day 1 and Day 3 of Part B at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post AZD1775 dose
  To assess the effect on QT interval corrected for heart rate (QTc) following multiple oral doses of AZD1775

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Terminal half-life for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Elimination rate constant for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Apparent clearance following oral administration for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Apparent volume of distribution for cocktail parent compounds (midazolam, omeprazole and caffeine) | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Area under the plasma concentration-time curve from zero to infinity for cocktail metabolites | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Area under the plasma concentration-time curve from time zero to the time "t" of the last quantifiable concentration for cocktail metabolites | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Time to reach maximum plasma concentration for cocktail metabolites | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Maximum plasma drug concentration for cocktail metabolites | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Terminal half-life for cocktail metabolites | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Elimination rate constant for cocktail metabolites | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Day 1, Part B Only: Area under the plasma concentration-time curve from time zero to 12 hours for AZD1775 | Blood samples are collected on Day 1 of Part B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 1, Part B only: Time to reach maximum plasma concentration for AZD1775 | Blood samples are collected on Day 1 of Part B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 1, Part B only: Maximum plasma drug concentration for AZD1775 | Blood samples are collected on Day 1 of Part B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 3, Parts A & B: Area under the plasma concentration-time curve from time zero to 12 hours for AZD1775 | Blood samples are collected on Day 3 of Part A and B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 3, Parts A & B: Time to reach maximum plasma concentration for AZD1775 | Blood samples are collected on Day 3 of Part A and B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 3, Parts A & B: Maximum plasma drug concentration for AZD1775 | Blood samples are collected on Day 3 of Part A and B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 3, Parts A & B: Minimum plasma drug concentration for AZD1775 | Blood samples are collected on Day 3 of Part A and B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 3, Parts A & B: Average concentration over a dosing interval for AZD1775 | Blood samples are collected on Day 3 of Part A and B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 3, Parts A & B: Apparent clearance at steady state for AZD1775 | Blood samples are collected on Day 3 of Part A and B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Day 3, Parts A & B: Fluctuation index (FI) over a dosing interval for AZD1775 | Blood samples are collected on Day 3 of Part A and B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Part B only: Accumulation ratio for area under the plasma concentration-time curve from time zero to twelve hours for AZD1775 | Blood samples are collected on Day 1 and 3 of Part B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
Part B only: Accumulation ratio for maximum plasma drug concentration for AZD1775 | Blood samples are collected on Day 1 and 3 of Part B at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of AZD1775 following single and multiple dose administration
dECG intervals (heart rate, RR, PR, QRS, QTcB, QTcF and QT) for absolute values and time-matched change from baseline | dECG intervals are performed on Day -1, Day 1, and Day 3 of Part B at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose
  To evaluate the effect of single and multiple doses of AZD1775 on cardiac (ECG) parameters
Changes in dECG morphology | dECG intervals are performed on Day -1, Day 1, and Day 3 of Part B at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose
  To evaluate the effect of single and multiple doses of AZD1775 on cardiac (ECG) parameters
Area under the plasma concentration-time curve from time zero to infinity ratios in relation to parent compound | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775
Maximum plasma drug concentration ratios in relation to parent compound | Blood samples are collected on Day -8, and Day 3 of Part A at pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose
  To describe the PK of midazolam, omeprazole and caffeine and their metabolites (1'-hydroxy-midazolam, 5-hydroxy-omeprazole, and paraxanthine) in the absence and presence of AZD1775

CONTACTS AND LOCATIONS:
Overall Officials: Lone Ottesen, MD, Study Director — AstraZeneca; Ding Wang, MD, Principal Investigator — Henry Ford Hospital
Locations (7):
- United States (7):
  - Research Site, Bingham Farms, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Lebanon, New Hampshire
  - Research Site, Cincinnati, Ohio
  - Research Site, Providence, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagard M, Ah-See ML, Strauss J, Wise-Draper T, Safran HP, Nadeau L, Edenfield WJ, Lewis LD, Ottesen LH, Li Y, Mugundu GM. Phase I study to assess the effect of adavosertib (AZD1775) on the pharmacokinetics of substrates of CYP1A2, CYP2C19, and CYP3A in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2023 Sep;92(3):193-203. doi: 10.1007/s00280-023-04554-3. Epub 2023 Jul 2. PMID 37394627
- [Derived] Nagard M, Ah-See ML, Strauss J, Wise-Draper T, Safran HP, Nadeau L, Edenfield WJ, Lewis LD, Rekic D, Dota C, Ottesen LH, Li Y, Mugundu GM. Adavosertib (AZD1775) does not prolong the QTc interval in patients with advanced solid tumors: a phase I open-label study. Cancer Chemother Pharmacol. 2023 Aug;92(2):141-150. doi: 10.1007/s00280-023-04555-2. Epub 2023 Jun 27. PMID 37368100